CLINICAL TRIAL: NCT04418973
Title: Analysis of Breath Volatile Organic Compounds After Dyspnea Induced in the Healthy Subject, by a Threshold Inspiratory Load and During a Maximal Breath Holding.
Brief Title: Analysis of Breath Volatile Organic Compounds After Dyspnea Induced in the Healthy Subject.
Acronym: Volatopnee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019_0074
Record Dates: First submitted 2020-02-12; First posted 2020-06-05 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Healthy Subjects
Keywords: Volatolom; Volatile organic compounds (VOCs); dyspnea; electronic nose; mass spectrometry
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - load/apnea (Experimental): Threshold inspiratory load then apnea
  Interventions: Other: VOCs analysis in exhaled air
- B- apnea/load (Experimental): apnea than threshold inspiratory load
  Interventions: Other: VOCs analysis in exhaled air

INTERVENTIONS:
Other: VOCs analysis in exhaled air — using an electronic nose and a mass spectrometry

SUMMARY:
The dyspnea is a common symptom in patients with many respiratory diseases particularly chronic obstructive airway diseases, but also cardiovascular pathologies, obesity, or also in the deconditioned healthy subjects.

Called volatolom corresponds to the set of volatile organic compounds (VOCs) contained in exhaled air.

The analysis of volatolom can be done either by the methods based on mass spectrometry which allows the identification of each VOC in the exhaled air or by the use of electronic noses which are more simple to use, less specific and produce a quantitive signal change based on pattern recognition algorithms providing a global profile of the VOC without identifying them.

The aim of the study is to determine whether the analysis of VOCs in exhaled air would identify biomarkers related to the intensity and type of experimental dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject
* no dyspnea
* non smoking or daily smoking more than 5 years packs
* perfect knowing of the French language
* the consent form signed
* affiliated to a health insurance plan

Exclusion Criteria:

* chronic disease
* history of asthma or Chronic obstructive pulmonary disease (COPD)
* personal or family atopy
* cannabis use
* electronic cigarette
* medication except contraception
* pregnant woman
* without liberty or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Comparison of variation of volatile organic compounds profiles in exhaled air during dyspnea and normal breathing. | at the only one study visit: around 2 hours
  Comparison of variation in VOC profiles in exhaled air of healthy subjects, over 2 types of dyspnea (inspiratory load and breath holding) relative to VOC profiles during normal rest ventilation. The VOC will be identified by their molecular mass (by the mass spectrometry) and the variations in the sensors properties of the electronic noses producing a quantitive signal change based on pattern recognition algorithms.

SECONDARY OUTCOMES:
Comparison of variation of volatile organic compounds profiles in exhaled air between the 2 types of dyspnea. | at the only one study visit: around 2 hours
  Comparison of variation of volatile organic compounds profiles in exhaled air between the 2 types of dyspnea (inspiratory load and breath holding).The VOC will be identified by their molecular mass (by the mass spectrometry) and the sensor deflection (by an electronic nose).
Correlation between the intensity of the affective component of the dyspnea and the variation of VOC profiles. | at the only one study visit: around 2 hours
  Correlation between the results of 2 questionnaires (affective multidimensional dyspnea and affective visual analogue scale) and the VOC profiles, in each of the 2 types of dyspnea.The VOC will be identified by their molecular mass (by the mass spectrometry) and the sensor deflection (by an electronic nose).
Correlation between the intensity of the sensory components of the dyspnea and the variation of VOC profiles. | at the only one study visit: around 2 hours
  Correlation between the results of 2 patient sensory questionnaires (sensory multidimensional dyspnea and sensory visual analogue scale) and the VOC profiles of dyspnea.The VOC will be identified by their molecular mass (by the mass spectrometry) and the sensor deflection (by an electronic nose).
Comparison of VOC profiles in exhaled air according to smoking status. | at the only one study visit: around 2 hours
  Comparison of VOC profiles in exhaled air of healthy subjects, in each of the 2 types of dyspnea smokers or non smokers. The VOC will be identified by their molecular mass (by the mass spectrometry) and the sensor deflection (by an electronic nose).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devillier, Principal Investigator — Hopital Foch
Locations (1):
- Foch hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No